CLINICAL TRIAL: NCT05424081
Title: The EMBER Trial for Weight Management Engagement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 19-422
Record Dates: First submitted 2022-06-10; First posted 2022-06-21 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Obesity
Keywords: obesity; weight loss; treatment engagement
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participant outcomes will be assessed by an outside company with no knowledge of randomization status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EMBER (Experimental): Self-help tool to increase weight management engagement
  Interventions: Behavioral: EMBER
- Control (Active Comparator): List of treatments
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: EMBER — Self-help tool to increase weight management engagement
  Arms: EMBER
Behavioral: Control — List of weight management programs
  Arms: Control

SUMMARY:
This study will test whether EMBER, a self-help tool to increase weight loss treatment engagement, helps veterans engage in Veterans Health Administration (VHA) weight management programs. Participants will be randomly assigned to receive EMBER or a list of weight management programs (the control group). They will answer questions about health beliefs and behaviors and share information from their medical record at the start of the study, 2-months after the start of the study, and 6-months after the start of the study. Participants will receive compensation for each of these contacts. Participants will also receive a reminder call 10 days after they enroll in the study. All study contacts will be over the phone. The main hypothesis is that people who receive EMBER will be more likely to use VHA weight management programs than people in the control group.

DETAILED DESCRIPTION:
Background Almost 40% of veterans using the Veterans Health Administration (VHA) have obesity. However, few patients use VHA's effective weight management programs. This study tests the effectiveness of EMBER, a self-directed tool with the goal of Enhancing Motivation for Better Engagement and Reach (EMBER) for weight management. It is available in paper and digital formats. EMBER is not a weight management program, instead it engages veterans in existing programs by informing and guiding choices about weight management.

Specific Aims

1. Assess whether veterans randomized to EMBER are more likely to have any weight management engagement at 2-month follow-up (per electronic medical record data supplemented with self-report) compared to those randomized to the control arm (information sheet listing available programs). (Primary Outcome)
2. Assess whether veterans randomized to EMBER have greater weight management program retention, weight management behaviors (e.g., physical activity), weight loss, and quality of life gains at 6-month follow-up compared to those randomized to the control arm. (Secondary Outcomes)
3. Assess factors likely to affect EMBER's implementation. Preliminary implementation outcomes will be assessed via RE-AIM (Reach, Effectiveness, Implementation) and the Proctor et al. implementation outcomes framework (Acceptability, Appropriateness, Costs, Fidelity). (Implementation Outcomes)

Methodology Randomized two site Hybrid Type 1 Effectiveness-Implementation Trial among veteran primary care patients with obesity in VA. Participants (N=470) will be randomized to EMBER or a control condition consisting of a list of available weight management programs. Logistic regressions will be used to assess Aims 1 and 2. Aim 3 results are descriptive.

ELIGIBILITY:
Inclusion Criteria:

* Veteran using primary care at VA Palo Alto or Houston in prior year
* BMI greater than or equal to 30 kg/m2

Exclusion Criteria:

* Age 80 or older
* Documentation of a suicide attempt in the past 30 days
* Hospitalization in the past 30 days
* Documentation or other evidence of cognitive impairment
* VA weight management program use in past 2 years
* Self-report from potential participant that they will not be in town for the majority of the 2 months following baseline
* Self-report from potential participant they plan to leave VA Palo Alto or Houston within the next 6 months
* Under age 18

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Weight management use | 2-months post randomization
  Dichotomous variable representing whether participant has 1+ VA weight management visits in the 2 months after baseline, per administrative data and/or self-report of use of VA weight management programs via single item question.

SECONDARY OUTCOMES:
Weight management use | 6-months post randomization
  Dichotomous variable representing whether participant has 1+ VA weight management visits in the 6 months after baseline, per administrative data and/or self-report of use of VA weight management programs via single item question.
Number of weight management visits | 6-months post-randomization
  Number of weight management program visits per administrative data.
New weight management behavior | 2- and 6-months post randomization
  Count of new weight management behaviors since baseline visit via self-report to question based on NHANES item assessing whether participant tried to lose weight and how. Lowest possible value 0 new weight management behaviors, no upper limit. Any change is considered meaningful.
Quality of life | 2- and 6-months post randomization
  Self-report of quality of life as assessed with the VR12 physical and mental health composite scores (Boston University School of Public Health). Scores are standardized T-scores with mean = 50 and a standard deviation of 10. For individuals on the physical health score, a 6.5 unit change is considering clinically meaningful. For individuals on the mental health score, a 7.9 unit change is considering clinically meaningful. At the population level, a 1 unit change is considered clinically meaningful.
Weight Loss | 6-months post randomization
  Based on difference between self-reported weight at baseline and 6-months, supplemented with medical record data when possible.
Physical Activity | 2- and 6-months post randomization
  Measured with L-Cat (Kiernen et al, 2013), which is a 6-level categorical measure. An increase of one category is a clinically meaningful difference.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Yelena Breland, PhD MS BA, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (2):
- United States (2):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be created and shared with qualified investigators.
Time Frame: Datasets will be available within 1 year of publication.
Access Criteria: Datasets meeting VA standards for disclosure to the public will be made available within 1 year of publication. Prior to distribution, a local privacy officer will certify that all datasets contains no PHI. Final data sets will be maintained locally until enterprise-level resources become available for long-term storage and access. Guidance on request and distribution processes will be provided by VA Office of Research & Development (ORD). Those requesting data will be asked to sign a Letter of Agreement.

REFERENCES:
- [Background] Breland JY, Fletcher TL, Maguen S, Timko C, Raikov I, Boothroyd DB, Frayne SM. The EMBER trial for weight management engagement: A hybrid type 1 randomized controlled trial protocol. Contemp Clin Trials. 2023 Dec;135:107364. doi: 10.1016/j.cct.2023.107364. Epub 2023 Oct 24. PMID 37884122

DOCUMENTS (1):
  • Informed Consent Form (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/81/NCT05424081/ICF_000.pdf